CLINICAL TRIAL: NCT02759939
Title: Right For Me: Birth Control Decisions Made Easier
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Responsible Party: Principal Investigator, Rachel L. Thompson, Assistant Professor, The Dartmouth Institute, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 00028721
Record Dates: First submitted 2016-02-03; First posted 2016-05-03 (Estimated); Results first posted 2019-11-19 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Contraception
Keywords: Shared Decision-Making; Patient-Provider Communication
MeSH Terms: interventions — Videotape Recording; Decision Support Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Experimental)
  Interventions: Other: Video + Prompt Card
- Arm 2 (Experimental)
  Interventions: Other: Decision Aids + Training
- Arm 3 (Experimental)
  Interventions: Other: Video + Prompt Card; Other: Decision Aids + Training
- Arm 4 (No Intervention)

INTERVENTIONS:
Other: Video + Prompt Card — 1. A brief video (available in English and Spanish) intended to be viewed by patients immediately before the health care visit. The video aims to enhance patients' motivation, skills, and self-efficacy to ask their health care providers three specific questions: (1) What are my options? (2) What are the pros and cons of those options? and (3) How likely are those pros and cons to happen to me?
  2. A prompt card (available in English and Spanish) intended to be provided to patients when they view the video and kept. The card aims to remind patients of the three questions presented in the video.
  Arms: Arm 1; Arm 3
Other: Decision Aids + Training — 1. Seven one-page decision aids on contraceptive methods (available in English and Spanish) intended to be used by health care providers with patients during the health care visit.
  2. A five-minute training video and accompanying written guidance (available in English) intended to be reviewed by health care providers before implementing the decision aids (and as frequently as desired thereafter). The training aims to enhance providers' motivation, skills, and self-efficacy to use the decision aids to facilitate shared decision-making in the health care visit.
  Arms: Arm 2; Arm 3

SUMMARY:
Right For Me is a study that aims to improve the conversations patients and health care providers have about birth control. Right For Me will test two different strategies for improving these conversations. The first strategy is to give patients a video to watch that encourages them to ask three specific questions in their health care visit, as well as a prompt card that reminds them of the three questions. The second strategy is to give health care providers a set of decision aids that describe available birth control methods, as well as training in how to use them with patients during the health care visit. Right For Me will test whether introducing one or both of these strategies leads to better conversations than providing health care as usual.

ELIGIBILITY:
Inclusion Criteria:

1. Completed a health care visit at a participating clinic
2. Assigned female sex at birth
3. Aged 15 to 49 years
4. Able to read and write English or Spanish
5. Not previously participated in the study

Exclusion Criteria:

1. Not completed a health care visit at a participating clinic (including a patient's parent or a person acting as a patient's legal proxy)
2. Not assigned female sex at birth
3. Aged under 15 or over 49 years
4. Unable to read and write English or Spanish
5. Previously participated in the study

Ages: 15 Years to 49 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 5038 (Actual)
Dates: Start 2016-07-01 (Actual); Primary Completion 2016-12-30 (Actual); Study Completion 2017-07-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rachel Thompson, PhD, Principal Investigator — Dartmouth College
Locations (1):
- The Dartmouth Institute for Health Policy and Clinical Practice, Lebanon, New Hampshire, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators will make an anonymized copy of the final participant-level data set and essential analysis syntax available to others for research purposes, either via data sharing on request or via digital repository deposition, before October 2018.

REFERENCES:
- [Background] Shepherd HL, Barratt A, Jones A, Bateson D, Carey K, Trevena LJ, McGeechan K, Del Mar CB, Butow PN, Epstein RM, Entwistle V, Weisberg E. Can consumers learn to ask three questions to improve shared decision making? A feasibility study of the ASK (AskShareKnow) Patient-Clinician Communication Model((R)) intervention in a primary health-care setting. Health Expect. 2016 Oct;19(5):1160-8. doi: 10.1111/hex.12409. Epub 2015 Sep 14. PMID 26364752
- [Background] Barr PJ, Thompson R, Walsh T, Grande SW, Ozanne EM, Elwyn G. The psychometric properties of CollaboRATE: a fast and frugal patient-reported measure of the shared decision-making process. J Med Internet Res. 2014 Jan 3;16(1):e2. doi: 10.2196/jmir.3085. PMID 24389354
- [Background] Elwyn G, Barr PJ, Grande SW, Thompson R, Walsh T, Ozanne EM. Developing CollaboRATE: a fast and frugal patient-reported measure of shared decision making in clinical encounters. Patient Educ Couns. 2013 Oct;93(1):102-7. doi: 10.1016/j.pec.2013.05.009. Epub 2013 Jun 12. PMID 23768763
- [Background] Weisman CS, Maccannon DS, Henderson JT, Shortridge E, Orso CL. Contraceptive counseling in managed care: preventing unintended pregnancy in adults. Womens Health Issues. 2002 Mar-Apr;12(2):79-95. doi: 10.1016/s1049-3867(01)00147-5. PMID 11879761
- [Background] Brehaut JC, O'Connor AM, Wood TJ, Hack TF, Siminoff L, Gordon E, Feldman-Stewart D. Validation of a decision regret scale. Med Decis Making. 2003 Jul-Aug;23(4):281-92. doi: 10.1177/0272989X03256005. PMID 12926578
- [Background] O'Connor, A. 1996. User Manual - Decision Regret Scale. Ottawa. Retrieved from http://decisionaid.ohri.ca/docs/develop/User_Manuals/UM_Regret_Scale.pdf
- [Background] Centers for Disease Control and Prevention. 2012. Pregnancy Risk Assessment Monitoring System (PRAMS) Phase 7 Questionnaire: Topic Reference. Atlanta, GA.
- [Background] Kavanaugh ML, Schwarz EB. Prospective assessment of pregnancy intentions using a single- versus a multi-item measure. Perspect Sex Reprod Health. 2009 Dec;41(4):238-43. doi: 10.1363/4123809. PMID 20444179
- [Derived] Thompson R, Manski R, Donnelly KZ, Stevens G, Agusti D, Banach M, Boardman MB, Brady P, Colon Bradt C, Foster T, Johnson DJ, Li Z, Norsigian J, Nothnagle M, Olson AL, Shepherd HL, Stern LF, Tosteson TD, Trevena L, Upadhya KK, Elwyn G. Right For Me: protocol for a cluster randomised trial of two interventions for facilitating shared decision-making about contraceptive methods. BMJ Open. 2017 Oct 22;7(10):e017830. doi: 10.1136/bmjopen-2017-017830. PMID 29061624
- See also: Study Website — http://www.rightforme.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The recruitment period was April 1, 2016 to December 30, 2016. Recruitment took place in 16 primary care and/or reproductive health care clinics in the Northeast United States.
Pre-assignment Details: This was a cluster randomized trial. The level of randomization was clinics.
Groups:
- Video + Prompt Card: A brief video intended to be viewed by patients in the clinic immediately before the health care visit that encouraged them to ask their providers three questions, and a small prompt card intended to remind them of the three questions presented in the video.
- Decision Aids + Training: A set of seven one-page decision aids on contraceptive methods intended to be used by providers with patients during the health care visit, as well as a brief training video and written guidance intended to be viewed by providers before beginning to use the decision aids (and as frequently as desired thereafter).
- Video + Prompt Card and Decision Aids + Training: A brief video intended to be viewed by patients in the clinic immediately before the health care visit that encouraged them to ask their providers three questions, and a small prompt card intended to remind them of the three questions presented in the video.
  And A set of seven one-page decision aids on contraceptive methods intended to be used by providers with patients during the health care visit, as well as a brief training video and written guidance intended to be viewed by providers before beginning to use the decision aids (and as frequently as desired thereafter).
- Usual Care: Care as usual.
Period: Overall Study
Arm/Group | Video + Prompt Card | Decision Aids + Training | Video + Prompt Card and Decision Aids + Training | Usual Care
Started (Represents participants who consented to the study and were eligible.) | 1256 | 1143 | 1393 | 1246
Analyzed at T1 (Participants with valid data on the item assessing occurrence of a conversation about contraception.) | 1245 | 1141 | 1388 | 1244
Eligible for T2 and T3 (We imposed additional eligibility criteria for the T2 and T3 surveys to minimize participant burden.) | 935 | 962 | 1022 | 853
Analyzed at T2 and/or T3 (Participants were not required to have completed the T2 survey to be eligible for the T3 survey.) | 303 | 278 | 373 | 304
Consented to T2 and T3 | 579 | 626 | 702 | 564
Completed | 200 | 171 | 239 | 203
Not Completed | 1056 | 972 | 1154 | 1043
Not completed — Missing data on first outcome assessed | 11 | 2 | 5 | 2
Not completed — Ineligible for T2 and T3 | 310 | 179 | 366 | 391
Not completed — Lost to Follow-up | 735 | 791 | 783 | 650

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Video + Prompt Card | Decision Aids + Training | Video + Prompt Card and Decision Aids + Training | Usual Care | Total
Number analyzed (Participants) | 1245 | 1141 | 1388 | 1244 | 5018
Age, Customized [Count of Participants; unit: Participants] — Source: Self-developed. Precise wording of item and response options is available on request.
  Participants
    15 to 19 years | 224 | 172 | 181 | 180 | 757
    20 to 24 years | 427 | 336 | 369 | 359 | 1491
    25 to 29 years | 341 | 299 | 336 | 290 | 1266
    30 to 34 years | 137 | 173 | 234 | 165 | 709
    35 to 39 years | 60 | 93 | 127 | 109 | 389
    40 to 44 years | 39 | 41 | 77 | 79 | 236
    45 to 49 years | 17 | 27 | 64 | 62 | 170
Sex: Female, Male [Count of Participants; unit: Participants] — Source: Self-developed. Precise wording of item and response options is available on request.
  Participants
    Female | 1245 | 1141 | 1388 | 1244 | 5018
    Male | 0 | 0 | 0 | 0 | 0
Current Gender Identity [Count of Participants; unit: Participants] — Source: Cahill et al., 2014. Precise wording of item and response options is available on request.
  Participants
    Female | 1224 | 1120 | 1370 | 1233 | 4947
    Male | 0 | 1 | 0 | 1 | 2
    Trans Woman | 0 | 0 | 0 | 0 | 0
    Trans Man | 4 | 2 | 4 | 1 | 11
    Genderqueer | 13 | 13 | 10 | 6 | 42
    Other | 2 | 0 | 1 | 2 | 5
    Two or more | 2 | 5 | 3 | 1 | 11
Ethnicity [Count of Participants; unit: Participants] — Source: US Census Bureau, 2015. Precise wording of item and response options is available on request.
  Participants
    Not of Hispanic, Latino, or Spanish origin | 1153 | 1085 | 1294 | 1080 | 4612
    Of Hispanic, Latino, or Spanish origin(s) | 71 | 44 | 63 | 145 | 323
    Missing | 21 | 12 | 31 | 19 | 83
Race [Count of Participants; unit: Participants] — Source: US Census Bureau, 2015. Precise wording of item and response options is available on request.
  Participants
    White | 991 | 1036 | 1238 | 1018 | 4283
    Black or African American | 49 | 12 | 27 | 70 | 158
    American Indian or Alaska Native | 11 | 9 | 10 | 12 | 42
    Asian | 93 | 15 | 15 | 16 | 139
    Native Hawaiian or Some other race(s) | 16 | 15 | 18 | 52 | 101
    Two or more | 62 | 43 | 53 | 54 | 212
    Missing | 23 | 11 | 27 | 22 | 83
Health literacy [Count of Participants; unit: Participants] — Source: Chew et al., 2008; Chew et al., 2004; Wallace et al., 2006; Dageforde et al., 2015; Sarkar et al., 2011. Precise wording of item and response options is available on request.
  Participants
    Limited | 264 | 221 | 296 | 280 | 1061
    Adequate | 964 | 912 | 1069 | 949 | 3894
    Missing | 17 | 8 | 23 | 15 | 63
Educational attainment [Count of Participants; unit: Participants] — Source: US Census Bureau, 2015. Precise wording of item and response options is available on request.
  Participants
    12th grade or less | 64 | 118 | 148 | 151 | 481
    High school graduate | 289 | 304 | 367 | 293 | 1253
    College or some college | 705 | 623 | 705 | 652 | 2685
    After Bachelor's degree | 169 | 88 | 145 | 130 | 532
    Missing | 18 | 8 | 23 | 18 | 67
Health insurance coverage [Count of Participants; unit: Participants] — Source: Jones et al., 2008. Precise wording of item and response options is available on request.
  Participants
    None | 212 | 206 | 231 | 98 | 747
    Temporary Medicaid | 21 | 33 | 24 | 22 | 100
    Medicaid | 186 | 296 | 465 | 526 | 1473
    Private | 650 | 491 | 526 | 481 | 2148
    Other | 136 | 84 | 105 | 88 | 413
    Two or more | 19 | 22 | 16 | 14 | 71
    Missing | 21 | 9 | 21 | 15 | 66
Survey language [Count of Participants; unit: Participants] — Source: Administrative data.
  Participants
    English | 1244 | 1140 | 1386 | 1219 | 4989
    Spanish | 1 | 1 | 2 | 25 | 29
Number of pregnancies [Count of Participants; unit: Participants] — Source: Self-developed. Precise wording of item and response options is available on request.
  Participants
    None | 800 | 496 | 715 | 663 | 2674
    One | 180 | 250 | 226 | 195 | 851
    Two | 99 | 175 | 180 | 150 | 604
    Three or more | 137 | 208 | 236 | 214 | 795
    Missing | 29 | 12 | 31 | 22 | 94
Number of births [Count of Participants; unit: Participants] — Source: Self-developed. Precise wording of item and response options is available on request.
  Participants
    None | 1008 | 732 | 875 | 804 | 3419
    One | 117 | 197 | 198 | 152 | 664
    Two | 63 | 128 | 185 | 154 | 530
    Three or more | 22 | 65 | 91 | 107 | 285
    Missing | 35 | 19 | 39 | 27 | 120
Number of abortions [Count of Participants; unit: Participants] — Source: Self-developed. Precise wording of item and response options is available on request.
  Participants
    None | 899 | 742 | 1086 | 981 | 3708
    One | 203 | 258 | 193 | 168 | 822
    Two | 82 | 89 | 59 | 47 | 277
    Three or more | 33 | 31 | 13 | 16 | 93
    Missing | 28 | 21 | 37 | 32 | 118
Number of miscarriages [Count of Participants; unit: Participants] — Source: Self-developed. Precise wording of item and response options is available on request.
  Participants
    None | 1124 | 943 | 1166 | 1029 | 4262
    One | 66 | 142 | 132 | 128 | 468
    Two | 10 | 27 | 30 | 43 | 110
    Three or more | 10 | 8 | 21 | 16 | 55
    Missing | 35 | 21 | 39 | 28 | 123
Previous contraceptive method(s) [Count of Participants; unit: Participants] — Operationalized as what, if any, contraceptive method(s) participants used in the 4 weeks before the health care visit. Source: Self-developed. Precise wording of item and response options is available on request.
  Participants
    Highly effective method(s) | 244 | 255 | 334 | 327 | 1160
    Less effective method(s) | 624 | 609 | 660 | 474 | 2367
    No methods | 162 | 187 | 154 | 164 | 667
    Missing | 4 | 1 | 6 | 4 | 15
    Not asked | 211 | 89 | 234 | 275 | 809

OUTCOME MEASURES:

1. Primary Outcome: Shared Decision-making About Contraceptive Methods
Description: Shared decision-making about contraceptive methods in the health care visit, measured using the three-item CollaboRATE measure (Barr et al., 2014; Elwyn et al., 2013). We used the version of CollaboRATE with a five-point response scale and adopted the binary scoring approach, which yields a score of 0 (no shared decision-making) and 1 (shared decision-making) for each participant. Note: 'pre-implementation participants' comprise those enrolled in the trial before clinics began implementing interventions and 'post-implementation participants' comprise those enrolled in the trial after clinics began implementing interventions (if relevant).
Time Frame: Immediately after the index health care visit (Time 1 (T1)) [for both pre-implementation and post-implementation participants]
Population: Participants with valid data on the primary outcome of shared decision-making about contraceptive methods and all covariates included in the adjusted analytic model. Data were collected at three time points from samples receiving care before (pre-implementation) and after (post-implementation) introduction of any intervention(s).
Measure: Count of Participants; unit: Participants
Arm/Group | Video + Prompt Card | Decision Aids + Training | Video + Prompt Card and Decision Aids + Training | Usual Care
Number analyzed (Participants) | 995 | 1031 | 1117 | 937
Participants
  Pre-implementation: number analyzed (Participants) | 296 | 414 | 345 | 299
  Pre-implementation: Shared decision-making | 165 | 272 | 222 | 190
  Pre-implementation: No shared decision-making | 131 | 142 | 123 | 109
  Post-implementation: number analyzed (Participants) | 699 | 617 | 772 | 638
  Post-implementation: Shared decision-making | 392 | 427 | 459 | 360
  Post-implementation: No shared decision-making | 307 | 190 | 313 | 278
Statistical Analysis 1: Comparison: Video + Prompt Card vs Usual Care; Test type: Superiority; p = 0.80, See below — Adjusted for multiple comparisons using the Scheffe method; Random effects logistic regression with a random intercept for clinic and adjustment for participant characteristics that differed across trial arms; Odds Ratio (OR) = 1.23
Statistical Analysis 2: Comparison: Decision Aids + Training vs Usual Care; Test type: Superiority; p = 0.32, See below — Adjusted for multiple comparisons using the Scheffe method; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 1.47
Statistical Analysis 3: Comparison: Video + Prompt Card vs Video + Prompt Card and Decision Aids + Training; Test type: Superiority; p = 0.99, See below — Adjusted for multiple comparisons using the Scheffe method; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.95
Statistical Analysis 4: Comparison: Decision Aids + Training vs Video + Prompt Card and Decision Aids + Training; Test type: Superiority; p = 0.72, See below — Adjusted for multiple comparisons using the Scheffe method; [statistical method as in outcome 1, analysis 1]; Odds Ratio (OR) = 0.80

2. Secondary Outcome: Conversation About Contraception
Description: Whether participants experienced a conversation about contraception in the health care visit, measured using a self-developed item. Note: 'pre-implementation participants' comprise those enrolled in the trial before clinics began implementing interventions and 'post-implementation participants' comprise those enrolled in the trial after clinics began implementing interventions (if relevant).
Time Frame: Immediately after the index health care visit (T1) [for both pre-implementation and post-implementation participants]
Reporting Status: Not Posted

3. Secondary Outcome: Satisfaction With Conversation About Contraception
Description: Participants' satisfaction with the conversation about contraception in the health care visit, measured using an adapted item (Weisman et al., 2002). Note: 'pre-implementation participants' comprise those enrolled in the trial before clinics began implementing interventions and 'post-implementation participants' comprise those enrolled in the trial after clinics began implementing interventions (if relevant).
Time Frame: Immediately after the index health care visit (T1) [for both pre-implementation and post-implementation participants]
Reporting Status: Not Posted

4. Secondary Outcome: Intended Contraceptive Method(s)
Description: What, if any, contraceptive method(s) participants intend to use in the next four weeks, measured using a self-developed checklist. Note: 'pre-implementation participants' comprise those enrolled in the trial before clinics began implementing interventions and 'post-implementation participants' comprise those enrolled in the trial after clinics began implementing interventions (if relevant).
Time Frame: Immediately after the index health care visit (T1) [for both pre-implementation and post-implementation participants]
Reporting Status: Not Posted

5. Secondary Outcome: Intention to Use a Highly Effective Contraceptive Method
Description: Whether participants intend to use at least one highly effective contraceptive method in the next four weeks, derived from data on intended contraceptive method(s). Note: 'pre-implementation participants' comprise those enrolled in the trial before clinics began implementing interventions and 'post-implementation participants' comprise those enrolled in the trial after clinics began implementing interventions (if relevant).
Time Frame: Immediately after the index health care visit (T1) [for both pre-implementation and post-implementation participants]
Reporting Status: Not Posted

6. Secondary Outcome: Values Concordance of Intended Contraceptive Method(s)
Description: Participants' perceptions of the degree of concordance between the contraceptive method(s) they intend(ed) to use and their individual values, needs, and preferences, measured using a self-developed item. Note: 'pre-implementation participants' comprise those enrolled in the trial before clinics began implementing interventions and 'post-implementation participants' comprise those enrolled in the trial after clinics began implementing interventions (if relevant).
Time Frame: Immediately after the index health care visit (T1); 4 weeks after the index health care visit (Time 2 (T2)); 6 months after the index health care visit (Time 3 (T3)) [for both pre-implementation and post-implementation participants]
Reporting Status: Not Posted

7. Secondary Outcome: Decision Regret About Intended Contraceptive Method(s)
Description: Participants' feelings of decision regret about the contraceptive method(s) they intended to use, measured using an adaptation of the five-item Decision Regret Scale (Brehaut et al., 2003; O'Connor, 1996). Note: 'pre-implementation participants' comprise those enrolled in the trial before clinics began implementing interventions and 'post-implementation participants' comprise those enrolled in the trial after clinics began implementing interventions (if relevant).
Time Frame: 4 weeks after the index health care visit (T2); 6 months after the index health care visit (T3) [for both pre-implementation and post-implementation participants]
Reporting Status: Not Posted

8. Secondary Outcome: Contraceptive Method(s) Used
Description: What, if any, contraceptive method(s) participants used in the last four weeks, measured using a self-developed checklist. Note: 'pre-implementation participants' comprise those enrolled in the trial before clinics began implementing interventions and 'post-implementation participants' comprise those enrolled in the trial after clinics began implementing interventions (if relevant).
Time Frame: as for outcome 7
Reporting Status: Not Posted

9. Secondary Outcome: Use of a Highly Effective Contraceptive Method
Description: Whether participants used at least one highly effective contraceptive method in the last four weeks, derived from data on contraceptive method(s) used. Note: 'pre-implementation participants' comprise those enrolled in the trial before clinics began implementing interventions and 'post-implementation participants' comprise those enrolled in the trial after clinics began implementing interventions (if relevant).
Time Frame: as for outcome 7
Reporting Status: Not Posted

10. Secondary Outcome: Use of Intended Contraceptive Method(s)
Description: Whether participants used their intended contraceptive method(s) in the last four weeks, derived from data on intended contraceptive method(s) and contraceptive method(s) used. Note: 'pre-implementation participants' comprise those enrolled in the trial before clinics began implementing interventions and 'post-implementation participants' comprise those enrolled in the trial after clinics began implementing interventions (if relevant).
Time Frame: as for outcome 7
Reporting Status: Not Posted

11. Secondary Outcome: Adherence to Contraceptive Method(s) Used
Description: Participants' adherence to the contraceptive method(s) they used in the last four weeks, measured using a self-developed, 21-item measure. Note: 'pre-implementation participants' comprise those enrolled in the trial before clinics began implementing interventions and 'post-implementation participants' comprise those enrolled in the trial after clinics began implementing interventions (if relevant).
Time Frame: as for outcome 7
Reporting Status: Not Posted

12. Secondary Outcome: Satisfaction With Contraceptive Method(s) Used
Description: Participants' satisfaction with the contraceptive method(s) they used in the last four weeks, measured using a self-developed item. Note: 'pre-implementation participants' comprise those enrolled in the trial before clinics began implementing interventions and 'post-implementation participants' comprise those enrolled in the trial after clinics began implementing interventions (if relevant).
Time Frame: as for outcome 7
Reporting Status: Not Posted

13. Secondary Outcome: Unintended Pregnancy (Pregnancy Timing Preferences)
Description: Participants' experience of one or more unintended pregnancies since the health care visit (as defined by their pregnancy timing preferences), measured using an adapted item (Centers for Disease Control and Prevention, 2012). Note: 'pre-implementation participants' comprise those enrolled in the trial before clinics began implementing interventions and 'post-implementation participants' comprise those enrolled in the trial after clinics began implementing interventions (if relevant).
Time Frame: 6 months after the index health care visit (T3) [for both pre-implementation and post-implementation participants]
Reporting Status: Not Posted

14. Secondary Outcome: Unintended Pregnancy (Pregnancy Seeking)
Description: Participants' experience of one or more unintended pregnancies since the health care visit (as defined by their pregnancy seeking), measured using an adapted item (Kavanaugh & Schwarz, 2009). Note: 'pre-implementation participants' comprise those enrolled in the trial before clinics began implementing interventions and 'post-implementation participants' comprise those enrolled in the trial after clinics began implementing interventions (if relevant).
Time Frame: 6 months after the index health care visit (T3) [for both pre-implementation and post-implementation participants]
Reporting Status: Not Posted

15. Secondary Outcome: Unwelcome Pregnancy
Description: Participants' experience of one or more unwelcome pregnancies since the health care visit, measured using an adapted item (Centers for Disease Control and Prevention, 2012). Note: 'pre-implementation participants' comprise those enrolled in the trial before clinics began implementing interventions and 'post-implementation participants' comprise those enrolled in the trial after clinics began implementing interventions (if relevant).
Time Frame: 6 months after the index health care visit (T3) [for both pre-implementation and post-implementation participants]
Reporting Status: Not Posted

16. Other Pre Specified Outcome: Exposure to Video
Description: Participants' exposure to the video and timing of exposure, measured using an adapted item (Shepherd et al., 2015). Note: 'pre-implementation participants' comprise those enrolled in the trial before clinics began implementing interventions and 'post-implementation participants' comprise those enrolled in the trial after clinics began implementing interventions (if relevant).
Time Frame: Immediately after the index health care visit (T1) [for both pre-implementation and post-implementation participants]
Reporting Status: Not Posted

17. Other Pre Specified Outcome: Exposure to Prompt Card
Description: Participants' exposure to the prompt card and timing of exposure, measured using a self-developed item. Note: 'pre-implementation participants' comprise those enrolled in the trial before clinics began implementing interventions and 'post-implementation participants' comprise those enrolled in the trial after clinics began implementing interventions (if relevant).
Time Frame: Immediately after the index health care visit (T1) [for both pre-implementation and post-implementation participants]
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Use of Three Questions
Description: Participants' use of each of the three patient questions in the health care visit, measured using three adapted items (Shepherd et al., 2015). Note: 'pre-implementation participants' comprise those enrolled in the trial before clinics began implementing interventions and 'post-implementation participants' comprise those enrolled in the trial after clinics began implementing interventions (if relevant).
Time Frame: Immediately after the index health care visit (T1) [for both pre-implementation and post-implementation participants]
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Exposure to Decision Aid(s)
Description: Participants' exposure to one or more of the decision aids and timing of exposure, measured using a self-developed item. Note: 'pre-implementation participants' comprise those enrolled in the trial before clinics began implementing interventions and 'post-implementation participants' comprise those enrolled in the trial after clinics began implementing interventions (if relevant).
Time Frame: Immediately after the index health care visit (T1) [for both pre-implementation and post-implementation participants]
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Acceptability of Video
Description: The acceptability of the video to participants, measured using a self-developed item. Note: 'pre-implementation participants' comprise those enrolled in the trial before clinics began implementing interventions and 'post-implementation participants' comprise those enrolled in the trial after clinics began implementing interventions (if relevant).
Time Frame: Immediately after the index health care visit (T1) [for both pre-implementation and post-implementation participants]
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Acceptability of Decision Aid(s)
Description: The acceptability of the decision aid(s) to participants, measured using a self-developed item. Note: 'pre-implementation participants' comprise those enrolled in the trial before clinics began implementing interventions and 'post-implementation participants' comprise those enrolled in the trial after clinics began implementing interventions (if relevant).
Time Frame: Immediately after the index health care visit (T1) [for both pre-implementation and post-implementation participants]
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: No adverse event data were collected.
Arm/Group | Video + Prompt Card | Decision Aids + Training | Video + Prompt Card and Decision Aids + Training | Usual Care
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0

LIMITATIONS AND CAVEATS:
Suboptimal retention at follow-up undermined our power to detect intervention effects on most secondary outcomes.

Modest rates of intervention implementation, according to patient-reported data, should be considered when results are interpreted.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes